

## SUPPLEMENTAL STATISTICAL ANALYSIS PLAN KTE-C19-106 TRANSLATIONAL ANALYSIS

| Sponsor: | Kite Pharma, Inc. |
|---|---|
| | 2400 Broadway |
| | Santa Monica, CA 90404 |
| | United States of America |
| <b>Product Name:</b> | KTE-C19 |
| Protocol: | A Phase 1-2 Multi-Center Study Evaluating the Safety and |
| | Efficacy of KTE-C19 in Combination with |
| | Atezolizumab in Subjects with Refractory Diffuse Large B- |
| | Cell Lymphoma (DLBCL) |
| NCT Number | NCT02926833 |
| Version Number: | Version 2.0 |
| Release Date: | 20 Feb 2020 |
| <b>Replaces Previous Version(s):</b> | Version 1.0; 04 March 2019 |

#### **CONFIDENTIALITY NOTICE**

This document contains confidential information of Kite Pharma Inc., a wholly owned subsidiary of Gilead Sciences Inc. This document must not be disclosed to anyone other than the site research staff and members of the Institutional Review Board/Independent Ethics Committee, a scientific review board or an equivalent. The information in this document cannot be used for any purpose other than the conduct of the clinical investigation without the prior written consent of Kite Pharma Inc. Questions regarding how this document should be used or the conduct of the clinical trial should be directed to the key sponsor contacts.

8.1.

## **TABLE OF CONTENTS**

| SUI | PLEM | ENTAL STATISTICAL ANALYSIS PLAN KTE-C19-106 | 1 |
|---|---|---|---|
| TAI | 3LE OF | CONTENTS | 2 |
| LIS | T OF T. | ABLES | 4 |
| LIS | T OF A | BBREVIATIONS | 5 |
| 1. | | ODUCTION | |
| 2. | | CTIVES | |
| ۷. | | | |
| | 2.1.<br>2.2. | Objectives | |
| 3. | FNDF | POINTS, SUBGROUPS AND COVARIATES | |
| ٥. | 3.1. | Biomarker datasets | |
| | 3.1. | Endpoints | |
| | 3.3. | Outcomes, Subgroups, and Covariates | |
| 4. | DEFI | NITIONS | 10 |
| | 4.1. | General | 10 |
| | 4.2. | Key Measurements of PD: Anti-CD19 CAR+ T-Cell | 10 |
| | 4.3. | Key Measurements of PD: Serum Cytokines | |
| | 4.4. | Key Measurements of CSF C-tables | |
| | 4.5.<br>4.6. | Key Measurements of CSF Cytokines | |
| | 4.0.<br>4.7. | Key Measurements of Atezolizumab | |
| | 4.8. | Key Measurements of Prognostic Marker PD-L1 | |
| 5. | ANAI | LYSIS SETS | 13 |
| | 5.1. | Modified Intent-to-treat Set (definition from Z6 clinical SAP 6.2) | 13 |
| | 5.2. | Safety Analysis Set (definition from clinical SAP 6.3) | |
| 6. | STAT | TSTICAL ANALYSIS | 14 |
| | 6.1. | General Methods | 14 |
| | 6.2. | Analysis | 15 |
| | | 6.2.1. Characterize the anti-CD19 CAR T cell expansion (PK) and serum | 1.0 |
| | | cytokine (PD) profile | 15 |
| | | | 7 |
| | | | , |
| 7. | REFE | D D | |
| | | | c |
| 8. | APPE | .IN | 0 |

| 8.2. | Analytic Visit Windows for PD Cytokines Key Measurement | 2 |
|------|---------------------------------------------------------|---|
| | Analytic Visit Windows for Atezolizumab PK | |
| | Analytic Visit Windows for Anti-KTE-C19 Antibody | |
| | CSF T-cell Analytes | |
| | Using Trapezoidal Rule to Approximate the AUC | |

## LIST OF TABLES

| Table 3-1. | Data overview on assay methods and biomarker lists | 8 |
|-------------|----------------------------------------------------|----|
| Table 6-1. | Non-parametric comparisons | |
| Table 8-1. | Cohort 1 visit window of PBMC in blood | |
| Table 8-2. | Cohort 2 visit window of PBMC in blood | 20 |
| Table 8-3. | Cohort 3 visit window of PBMC in blood | 20 |
| Table 8-4. | Phase 2 visit window of PBMC in blood | 20 |
| Table 8-5. | Cohort 1 visit window of PD cytokines | 22 |
| Table 8-6. | Cohort 2 visit window of PD cytokines | |
| Table 8-7. | Cohort 3 visit window of PD cytokines | |
| Table 8-8. | Atezo PK visit window | |
| Table 8-9. | Atezo ATA visit window | 23 |
| Table 8-10. | Anti-KTE-C19 antibody visit window | |
| Table 8-11. | CSF T-cell analytes | |

#### LIST OF ABBREVIATIONS

Atezo Atezolizumab
AE Adverse event

ASCT Autologous stem cell transplant

ATA Anti-tumor activity
AUC Area under the curve

Axicabtagene ciloleucel / Autologous T cells transduced with retroviral vector containing anti-CD19

KTE-C19 CD28/CD3 zeta chimeric antigen receptor

CAR Chimeric antigen receptor

CR Complete response / Complete remission

CRS Cytokine release syndrome

CSF Cerebrospinal fluid

DLBCL Diffuse large B cell lymphoma

IHC Immunohistochemistry

LYMLE Lymphocytes/Leukocytes (%)

mITT Modified intent-to-treat

MONOLE Monocytes/Leukocytes (%)

NE Neurotoxicity event

NHL Non-Hodgkin Lymphoma

PBMC Peripheral blood mononuclear cells

PD Progressive disease

PK/PD Pharmacokinetic / Pharmacodynamic
PMBCL Primary mediastinal B cell lymphoma
PR Partial response / Partial remission
RCR Replication competent retrovirus

SAE Serious adverse event

SD Stable disease

SOA Schedule of assessments

Study day 0 The first day that axicabtagene ciloleucel is administered to the subject

WBC White Blood Cell or Leukocytes

## 1. INTRODUCTION

This supplemental statistical analysis plan outlines the analyses of PK/PD, product characteristics, and other biomarkers in support of the regulatory filling for KTE-C19 in combination with Atezolizumab in subjects with refractory DLBCL. The analysis will be conducted for biomarker data within protocol KTE-C19-106 (ZUMA-6), amendment 1 dated 21 Sep 2017.

# 2. OBJECTIVES

# 2.1. Objectives

• Characterize the anti-CD19 CAR T cell expansion (PK) and serum cytokine (PD) profile



•



•



• Characterize the expression of CD19 target and PD-L1 expression in tumor biopsies at baseline, post treatment and at relapse; comparative analysis between Zuma 6 and Zuma 1

# 2.2. Hypothesis



# 3. ENDPOINTS, SUBGROUPS AND COVARIATES

## 3.1. Biomarker datasets

Table 3-1. Data overview on assay methods and biomarker lists

| Data type | Assay method/Sample type | Biomarker set |
|---|---|---|
| PK data (CAR<br>T) | qPCR/PBMC | number of CAR T cells (/µL), %PBMC |
| PK data<br>(Atezo) | Immunoassays/serum samples | <ul><li>Anti-Atezo Antibody</li><li>Atezo concentrations (ng/mL)</li></ul> |
| PD data<br>(cytokines) | Cytokine assay/serum sample | • Pro-inflammatory and immune modulating cytokines: IL-6 (pg/mL), TNFα (pg/mL), IL-10 (pg/mL), IL-2 (pg/mL), GM-CSF (pg/mL), IL 15 (pg/mL), IL-17 (pg/mL), IFNγ (pg/mL), IL-12p40/p70 (pg/mL); |
| | | Immune effector molecules: Granzyme A (pg/mL), B (pg/mL), Perforin (pg/mL) |
| | | • Correlates of acute phase response: CRP (mg/mL), Ferritin (pg/mL), sIL-2Ra (pg/mL) |
| | | • Chemokines: MIP-1α (pg/mL), MIP-1β (pg/mL), IP-10 (pg/mL), MCP-4 (pg/mL) |
| CSF cytokines | Cytokine assay/CSF sample | Biomarker list are the same with those in the PD cytokines |
| CSF T-cell | PCR complemented by Flow cytometry/CSF sample | Analytes are listed in Appendix 8.5 |
| PD-L1 and<br>CD19 IHC, in<br>addition to<br>other B cell<br>markers<br>(CD20, PAX5,<br>CAR T cell<br>presence) | Immunohistochemistry (IHC) and gene expression profiling / Fresh tumor biopsies (NeoGenomics) | <ul><li>PD-L1: H Score</li><li>CD 19</li></ul> |

## 3.2. Endpoints

All definitions are generally applied to PK/PD.

- Analyte baseline is defined as the last value measured prior to conditioning chemotherapy.
  - Other analytes at baseline include CD-19 H score and Baseline Tumor Burden.
- Change from baseline at Day X is defined as the difference of the value at Day X and at the baseline. i.e. Analyte level at Day X Analyte level at Baseline
- Fold change from baseline at Day X is defined as:

Analyte level at Day X

Analyte level at Baseline

- **Peak of analyte post KTE-C19 infusion** is defined as the maximum level measured post infusion.
- Time to peak post KTE-C19 infusion is defined as "Peak Date Dosing Date + 1".
- Area-Under-Curve (AUC) measures the total level of analyte overtime and is defined as the area under the curve in an analyte profile plot against scheduled visits as specified for each analyte.
- **PD-L1 expression** {Bot 2015, Chen 2013} is an expression level of PD-L1 on tumor tissue evaluated using a continuous value of H score derived by % cells expressing PD-L1 times intensity of expression.

#### 3.3. Outcomes, Subgroups, and Covariates

- Responder (PR/CR) vs Non-responder (Others)
- The worst neurotoxicity grade was "Grade 3 or higher (NEG3+)" vs. Others (NEG2)
- The worst neurotoxicity grade was "Grade 2 or higher (NEG2+)" vs. Others (NEG1)
- The worst CRS grade was "Grade 3 or higher" (CRSG3+) vs. Others (CRSG2)
- The worst CRS grade was "Grade 2 or higher" (CRSG2+) vs. Others (CRSG1)
- Best response: Complete Response (CR) vs. Partial Response (PR) vs. Non-responders
- Baseline covariates will be utilized if appropriate (list of baseline covariates refer to clinical SAP)

#### 4. **DEFINITIONS**

#### 4.1. General

**Study day 0** is defined as the day the subject received the first KTE-C19 infusion. The day prior to study day 0 will be study day -1. Any days after enrollment and prior to study day -1 will be sequential and negative integer-valued.

**Baseline** is defined as the last non-missing value measured on or prior to conditioning chemotherapy.

**Baseline of retreatment** is the last record on or prior to conditioning chemotherapy retreatment if the subject is eligible for retreatment with axicabtagene ciloleucel.

**KTE-C19 treatment period** begins on the day of the first KTE-C19 infusion up through and including 30 days after the KTE-C19 infusion.

## 4.2. Key Measurements of PD: Anti-CD19 CAR+ T-Cell

The expansion and persistence of anti-CD19 CAR T cells in peripheral blood will be monitored by qPCR analysis.

#### Scheduled blood draw for anti-CD19 CAR T cell

This SSAP will focus on the anti-CD19 CAR T cell data collected as per planned assessment. The schedule of assessments and the analytic visit windows are defined in Appendix 8.1.

#### Number of CAR T (cells/ µL blood) is defined as:

White Blood Cell counts × (Monocytes (%) + Lymphocytes (%)) × CAR<sup>+</sup>PBMCs (%)

**Peak of CAR T cell (cells/ \muL blood)** is defined as the maximum absolute number of CAR T cells in serum attained after Day 0.

**Time-to-Peak of CAR T cell (days)** is defined as "Peak Date – Dosing Date + 1".

Area-Under-Curve (AUC) of level of CAR T cell (cells/ μL • days) is defined as the area under the curve in a plot of levels of CAR T cells against scheduled visits. For Zuma 6 Cohort 1: From Day 0 to Day 28, For Zuma 6 Cohort 2 and 3: From Day 0 to Day 35. This AUC measures the total levels of CAR T cells overtime. Given the CAR+ T cell are measured at certain discrete time points, the trapezoidal rule will be used to estimate the AUCs.

**CAR T PEAK/Tumor burden:** ratio of CAR T Peak and baseline tumor burden local (investigator's assessment) will be assessed.

PK anlaytes (nCART, nCAR T Peak, or nCAR T AUC)

Baseline Tumor Burden (SPD) (mm^2) from local lab

## 4.3. Key Measurements of PD: Serum Cytokines

**Scheduled blood draw for cytokines:** Within approximately 5 days of eligibility confirmation (Enrollment/Leukapheresis) as baseline, Day 0, Day 3, Day 7, and on day of discharge of hospitalization, Week 2 (Day 14) ( $\pm$  2 days), and Week 4 (Day 28) ( $\pm$  2 days). This SSAP will focus on the cytokine data collected from baseline to Day 28. The SOA and analytic visit window is defined in Appendix 8.2.

**Baseline of cytokines** is defined as the last value measured prior to conditioning chemotherapy.

Fold change from baseline at Day X is defined as

Cytokine level at Day X — Cytokine level at Baseline
Cytokine level at Baseline

**Peak of cytokine post baseline** is defined as the maximum level of cytokine in serum attained after baseline up to Day 28.

**Time to peak of cytokine post KTE-C19 infusion** is defined as "Peak Date – Dosing Date + 1".

**Area-Under-Curve (AUC) of cytokine levels from baseline to Day 28**: is defined as the area under the curve in a plot of levels of cytokine against scheduled visits from baseline to Day 28. This AUC measures the total levels of cytokine overtime. Given the cytokine and CAR+ T cell are measured at certain discrete time points, the trapezoidal rule will be used to estimate the AUCs.

#### 4.4. Key Measurements of CSF T-cells



## 4.5. Key Measurements of CSF Cytokines

CSF cytokines are similar to those in the PD cytokines.

CSF sample collection has no scheduled assessment visits. Peak and AUC analysis are not applied to CSF cytokines.

4.



4.7

•

• Serum Atezolizumab concentration (ng/mL)

Serum samples will be assayed for atezolizumab concentrations using validated immunoassay {Fehrenbacher 2016}.

**Scheduled blood draw for Atezolizumab:** Refer to Appendix 8.3 for detailed information.

## 4.8. Key Measurements of Prognostic Marker PD-L1

PD-1 is an activation/exhaustion marker of cytolytic T cells and its expression is upregulated on the surface of CAR T cells beginning prior to infusion and is further enhanced during in vitro exposure to CD19-expressing target cells {Bot 2015, Herbst 2014}. PD-1 surface expression is also increased following CAR T cell infusion {Perez 2015}. The following key measurements will be analyzed for PD-L1 marker:

**H score** = % cell expressing PD-L1 x intensity of expression

## 5. ANALYSIS SETS

## 5.1. Modified Intent-to-treat Set (definition from Z6 clinical SAP 6.2)

The mITT set will consist of all subjects enrolled and treated with the target dose of axicabtagene ciloleucel at  $2 \times 10^6$  CAR T cells/kg ( $1.0 \times 10^6$  anti-CD19 CAR T cells/kg to  $2.4 \times 10^6$  anti-CD19 CAR T cells/kg) and at least 1 dose of atezolizumab as determined upon completion of Phase 1 and Phase 2 portions of the study.

## 5.2. Safety Analysis Set (definition from clinical SAP 6.3)

The safety analysis set (SAS) is defined as all subjects treated with any dose of axicabtagene ciloleucel.

#### 6. STATISTICAL ANALYSIS

#### **6.1.** General Methods

The following methods will be applied to the data analysis when applicable.

• Summary statistics will summarize data in frequency (N, %) and quartile range (Minimum, 1 quartile (Q1), Median, 3 quartile (Q3), Maximum) in overall and by appropriate subgroups and covariates (Section 3.3).



#### • Logistic Regression for binary outcomes

Binary outcome implies there are only two possible outcomes to a certain situation. Logistic regression will be conducted to describe and explain the relationship between an explanatory variable (predictor) and an outcome variable {Hosmer 2013}. Number of evaluable subjects for each group, Odds Ratio with 95% Confidence Interval, and raw unadjusted p value will be reported. Predictive probability will be plotted.

## • Nominal Logistic Regression for categorical outcomes

The categorical outcome has a limited number of possible outcomes. Nominal logistic regression {Hosmer 2013} will be used to describe and explain the relationship between an



comparison followed by pairwise comparisons using Dunn's test with Holm's adjustment method {Dunn 1964} implemented in the 'dunn.test' package for R {Dinno 2015}.

## 6.2. Analysis

# 6.2.1. Characterize the anti-CD19 CAR T cell expansion (PK) and serum cytokine (PD) profile

- Safety analysis set will be used for an overall PK/PD profile
- PK/PD profile overtime will be analyzed using summary statistics described in Section 6.1
- Comparison of PK/PD by subgroups will be conducted for special population, subgroups by baseline covariates (in Section 3.3) and safety and efficacy
  - Wilcoxon rank sum test will be used to compare the PK/PD profiles among the subgroups. See Table 6-1 for details.
  - For comparisons among CR vs PR vs Non-responders, Kruskal-Wallis test will be conducted. Further pairwise comparisons among these three groups, following a significant Kruskal-Wallis test, will be using Dunn's test with Holm's adjustment method.
- The Median Line plot with interquartile range (IQR) will be produced for overall cohort or by subgroups.

Table 6-1. Non-parametric comparisons

| | | | Key Measu | irements |
|---|---|---|---|---|
| Covariate | Subgroups | Method | CAR T Cell<br>Expansion in Blood | Cytokine Levels<br>in Serum |
| Response | Responder vs Non-<br>responder | Wilcoxon rank sum test | | |
| Worst<br>Neurotoxicity | Grade 3 or higher vs. grade 2 or lower | Wilcoxon rank sum test | | |
| Worst<br>Neurotoxicity | Grade 2 or higher vs. grade 1 or lower | Wilcoxon rank sum test | • AUC | • AUC |
| Worst CRS | Grade 3 or higher vs. grade 2 or lower | Wilcoxon rank sum test | • Peak | • Peak |
| Worst CRS | Grade 2 or higher vs. grade 1 or lower | Wilcoxon rank sum test | | |
| Best response | Complete Response vs. Partial Response vs. Non-responders | Kruskal-Wallis test | | |



## subjects

- Atezo PK will be summarized with summary statistics (Section 6.1) overtime and compared at selected Atezo dosing time
- Comparison of Atezo PK will be conducted for special population or subgroups by baseline covariates (in Section 3.3)
- Comparison of Atezo PK will be conducted by safety and efficacy subgroups

# **6.2.5.** Characterize the products

• Safety analysis set will be used for analysis



#### 7. REFERENCES

- Bot A, Kochenderfer J, Mardiros A, Perez A, Navale L, Chang R, et al. Biomarker analysis of patients treated with anti-CD19 chimeric antigen receptor (CAR) T cells.

  American Society of Clinical Oncology (ASCO) Annual Meeting 2015; Abstract #3028.
- Chen BJ, Chapuy B, Ouyang J, Sun HH, Roemer MG, Xu ML, et al. PD-L1 expression is characteristic of a subset of aggressive B-cell lymphomas and virus-associated malignancies. Clin Cancer Res 2013;19 (13):3462-73.
- Dinno A. Nonparametric Pairwise Multiple Comparisons in Independent Groups using Dunn's Test. Stata Journal 2015;15 (1):292-300.
- Dunn OJ. Multiple Comparisons Using Rank Sums. Technometrics 1964;6 (3):241-52.
- Fehrenbacher L, Spira A, Ballinger M, Kowanetz M, Vansteenkiste J, Mazieres J, et al. Atezolizumab versus docetaxel for patients with previously treated non-small-cell lung cancer (POPLAR): a multicentre, open-label, phase 2 randomised controlled trial. Lancet 2016;387 (10030):1837-46.
- Gelman A, Hill J. Linear regression. In: Gelman A, Hill J, eds. Data Analysis Using Regression and Multilevel/Hierarchical Models. 5th ed. New York: Cambridge University Press; 2006: 31-77.
- Herbst RS, Soria JC, Kowanetz M, Fine GD, Hamid O, Gordon MS, et al. Predictive correlates of response to the anti-PD-L1 antibody MPDL3280A in cancer patients. Nature 2014;515 (7528):563-7.
- Holm S. A Simple Sequentially Rejective Multiple Test Procedure. Scandinavian Journal of Statistics 1979;6 (2):65-70.
- Hommel G. A Stagewise Rejective Multiple Test Procedure Based on a Modified Bonferroni Test. Biometrika 1988;75 (2):383-6.
- Hosmer DW, Lemeshow S, Studivant RX. Introduction to the Logistic Regression Model. In: Balding DJ, Cressie NAC, Fitzmaurice GM, eds. Applied Logistic Regression. 3rd ed. Hoboken, New Jersey: John Wiley & Sons, Inc.; 2013: 1-47.
- Kruskal WH, Wallis WA. Use of Ranks in One-Criterion Variance Analysis. Journal of the American Statistical Association 1952;47 (260):583-621.
- Perez A, Navale L, Rossi JM, Shen Y-w, Jiang Y, Sherman M, et al. Pharmacodynamic Profile and Clinical Response in Patients with B-Cell Malignancies of Anti-CD19 CAR T-Cell Therapy. Blood 2015;126 (23):2042.

Siegel S. The One-Sample Runs Test. In: Morgan CT, ed. Nonparametric Statistics: For the Behavioral Sciences. New York: McGraw-Hill Book Company, Inc.; 1956: 75-83.

Wilcoxon F. Individual Comparisons by Ranking Methods. Biometrics Bulletin 1945;1 (6):80-3.

## 8. APPENDIX

## 8.1. Analytic Visit Windows for CAR T Cells in Blood

#### Table 8-1. Cohort 1 visit window of PBMC in blood

| Analytic<br>Visit | Baseline | Day<br>0 | Day 7 | Day 14 | Day 21 | Day 28 | Day 42 | Day 49 | Day 63 | Day 70 | Day 84 | Day 91 | | | Month 9<br>Day 270 | 12 Day | MONTH<br>15 Day<br>450 | 18 Day | MONTH<br>24 Day<br>720 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Target Day | Baseline | 0 | 1 - 7 | $14 \pm 2$ | $21 \pm 2$ | $28 \pm 2$ | 42 ± 2 | 49 ± 2 | $63 \pm 2$ | $70 \pm 2$ | $84 \pm 2$ | 91 ± 2 | $114\pm7$ | | | | | | |
| Lab Window | <=-5 | [,] | [1, 10] | [11, 17] | [18, 24] | [25, 35] | [36, 45] | [46, 56] | [57, 66] | [67, 77] | [78, 87] | [88, 102] | [103, 147] | [148, 225] | [226, 315] | [316, 405] | [406, 495] | [496, 585] | [> 586] |

## Table 8-2. Cohort 2 visit window of PBMC in blood

| Analytic<br>Visit | Baseline | Day<br>0 | Day 7 | Day 14 | Day 17 | Day 21 | Day 35 | Day 42 | Day 56 | Day 63 | Day 77 | Day 84 | | Month 6<br>Day 180 | | | MONTH<br>15 Day<br>450 | 18 Day | MONTH<br>24 Day<br>720 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Target Day | Baseline | 0 | 7 | 14 ± 2 | $17 \pm 2$ | $21 \pm 2$ | $35 \pm 2$ | $42 \pm 2$ | $56 \pm 2$ | $63 \pm 2$ | $77 \pm 2$ | $84 \pm 2$ | $107 \pm 7$ | | | | | | |
| Lab Window | v <= -5 | [,] | [1, 10] | [11, 15] | [16, 18] | [19, 28] | [29, 38] | [39, 49] | [50, 59] | [60, 70] | [71, 80] | [81, 95] | [96, 143] | [144, 225] | [226, 315] | [316, 405] | [406, 495] | [496, 585] | [> 586] |

#### Table 8-3. Cohort 3 visit window of PBMC in blood

| Analytic<br>Visit | Baseline | Day<br>0 | Day 7 | Day 14 | Day 22 | Day 35 | Day 43 | Day 49 | Day 64 | Day 69 | | Month 6<br>Day 180 | Month 9 Day<br>270 | | | | MONTH 24<br>Day 720 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Target Day | Baseline | 0 | 1 - 7 | $14 \pm 2$ | $22 \pm 2$ | $35 \pm 2$ | $43 \pm 2$ | $49 \pm 2$ | $64 \pm 2$ | $69 \pm 2$ | 94 ± 7 | | | | | | |
| Lab Window | <=-5 | [,] | [1, 10] | [11, 17] | [18, 28] | [29, 38] | [39, 45] | [46, 56] | [57, 66] | [67, 77] | [78, 143] | [144, 225] | [226, 315] | [316, 405] | [406, 495] | [496, 585] | [> 586] |

## Table 8-4. Phase 2 visit window of PBMC in blood

| Analytic<br>Visit | Baseline | Day<br>0 | Day<br>3 | , , | W2<br>Day 14 | | Day 28 | Day 42 | Day 49 | Day 63 | Day 70 | | | | Month 12<br>Day 360 | 15 Day | | | Month 36<br>Day 1080 | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Target Day | Baseline | 0 | | | 14 ± 2 | $22 \pm 2$ | $28 \pm 2$ | $43 \pm 2$ | $49 \pm 2$ | $64 \pm 2$ | $69 \pm 2$ | 94 ± 2 | | | | | | | | | |
| Lab<br>Window | <=-5 | [,] | [2, 4] | [5, 10] | [11, 17] | [18, 25] | [26, 35] | [36, 45] | [46, 56] | [57, 66] | [67, 77] | [78, 143] | [144, 225] | [226, 315] | [316, 405] | [406, 495] | [496, 585] | [586,900<br>] | [901, 1260] | [1261,<br>1620] | [>1621, ] |

- PBMCs Blood draw for PBMCs include the analysis of lymphocytes prior to axicabtagene ciloleucel infusion and lymphocytes, anti KTE-C19 CAR T cells, and RCR after CAR T infusion.
- Baseline is at enrollment and before leukapheresis.

CONFIDENTIAL Page 21

## 8.2. Analytic Visit Windows for PD Cytokines Key Measurement

## Table 8-5. Cohort 1 visit window of PD cytokines

| Analytic Visit | Baseline | Day 0 | Day 1 | Day 4 | Day 7 | Day 14 | Day 21 | Day 28 | Day 42 | Day 49 | Day 70 | Day 91 | | Month 6<br>Day180 | | 12 Day | 15 Day | | MONTH 24<br>Day 720 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Target Day | Baseline | 0 | 1 | 4 | 7 | $14 \pm 2$ | $21 \pm 2$ | $28 \pm 2$ | $42 \pm 2$ | $49 \pm 2$ | $70 \pm 2$ | $91 \pm 2$ | $114 \pm 7$ | | | | | | |
| Lab Window | <=-5 | [0,0] | [1,2] | [3,5] | [6, 10] | [11, 17] | [18, 24] | [25, 35] | [36, 45] | [46, 63] | [64, 84] | [85, 102] | [103, 147] | [148, 225] | [226, 315] | [316, 405] | [406, 495] | [496, 585] | [> 586] |

## Table 8-6. Cohort 2 visit window of PD cytokines

| Analytic<br>Visit | Baseline | Day 0 | Day 1 | Day 4 | Day 7 | Day 14 | Day 21 | Day 35 | Day 42 | Day 63 | Day 84 | | Month 6<br>Day 180 | | | | MONTH 18<br>Day 540 | MONTH 24<br>Day 720 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Target Day | Baseline | 0 | 1 | 4 | 7 | $17 \pm 2$ | 21 ± 2 | $35 \pm 2$ | 42 ± 2 | $63 \pm 2$ | 84 ± 2 | $107 \pm 7$ | | | | | | |
| Lab Window | v <= -5 | [0, 0] | [1, 2] | [3, 5] | [6, 10] | [11, 17] | [18, 28] | [29, 38] | [39, 56] | [57, 77] | [78, 95] | [96, 147] | [148, 225] | [226, 315] | [316, 405] | [406, 495] | [496, 585] | [> 586] |

# Table 8-7. Cohort 3 visit window of PD cytokines

| Analytic<br>Visit | Baseline | Day 0 | Day 1 | Day 4 | Day 7 | Day 14 | Day 22 | Day 35 | Day 49 | Day 69 | Day 94 | Month 6 Day<br>180 | Month 9 Day<br>270 | MONTH 12<br>Day 360 | MONTH 15<br>Day 450 | | MONTH 24<br>Day 720 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Target Day | Baseline | 0 | 1 | 4 | 7 | $14 \pm 2$ | $22 \pm 2$ | 35 ± 2 | 49 ± 2 | $69 \pm 2$ | 94 ± 7 | | | | | | |
| Lab Window | v < = -5 | [0, 0] | [1, 2] | [3, 5] | [6, 10] | [11, 17] | [18, 28] | [29, 38] | [46, 56] | [67, 77] | [78, 143] | [144, 225] | [226, 315] | [316, 405] | [406, 495] | [496, 585] | [> 586] |

• Baseline is at enrollment and before leukapheresis.

## 8.3. Analytic Visit Windows for Atezolizumab PK

Table 8-8. Atezo PK visit window

| | Analytic Visit | Day21 Pre | Day 21 Post | Day 42 | Day 63 | Day 84 | Day 174 |
|---|---|---|---|---|---|---|---|
| Phase1<br>Cohort1 | Target Day | 21 ± 2 | 21 ± 2 | 42 ± 2 | 63 ± 2 | 84 ± 2 | |
| | Proposed Window | [17, 31] | [17, 31] | [32, 52] | [53,73] | [74, 94] | [95, ] |
| D) 4 | Analytic Visit | Day 14 Pre | Day 14 Post | Day 35 | Day 56 | Day 77 | Day 167 |
| Phase1<br>Cohort2 | Target Day | 14 ± 2 | 14 ± 2 | 35 ± 2 | 56 ± 2 | $77 \pm 2$ | |
| | Proposed Window | [10, 24] | [10, 24] | [25, 45] | [46, 66] | [67, 87] | [88, ] |
| Phase1<br>Cohort3 &<br>Phase 2 | Analytic Visit | Day 1 Pre | Day 1 Post | Day 22 | Day 43 | Day 64 | Day 154 |
| | Target Day | 1 | 1 | $22 \pm 2$ | 43 ± 2 | $64 \pm 2$ | |
| | Proposed Window | [1, 10] | [1, 10] | [11, 32] | [33, 53] | [54, 74] | [75, ] |

Table 8-9. Atezo ATA visit window

| Cohort 1 | Analytic Visit | Day 21 <sup>B</sup> | Day 42 <sup>A</sup> | Day 63 <sup>A</sup> | Day 84 <sup>B</sup> |
|---|---|---|---|---|---|
| | Target Day | 21 ± 2 | 42 ± 2 | 63 ± 2 | 84 ± 2 |
| | Lab Window | [,] | [,] | [,] | [,] |
| Cohort 2 | Analytic Visit | Day 14 <sup>B</sup> | Day 35 <sup>A</sup> | Day 56 <sup>A</sup> | Day 77 <sup>B</sup> |
| | Target Day | 14 ± 2 | 35 ± 2 | 56 ± 2 | 77 ± 2 |
| | Lab Window | [,] | [,] | [,] | [, ] |
| Cohort 3 | Analytic Visit | Day 1 <sup>B</sup> | Day 22 <sup>A</sup> | Day 43 <sup>A</sup> | Day 64 <sup>B</sup> |
| | Target Day | 1 | 22 ± 2 | 43 ± 2 | 64 ± 2 |
| | Lab Window | [,] | [,] | [, ] | [,] |

#### Notes:

Long-term follow-up period: Take a single time point sample  $\geq 90$  days after the last atezolizumab infusion for the initial course of therapy and another single time point sample after the retreatment period (if applicable).

Take a sample prior to the atezolizumab infusion for the initial course of treatment and during the retreatment period (if applicable). For the initial course of treatment only, take a sample at  $30 \text{ min } \pm 10 \text{ min } \pm 1$ 

Take sample prior to the atezolizumab infusion. This sample is NOT required during the retreatment period.

Take sample prior to the atezolizumab infusion for the initial course of treatment and during the retreatment period (if applicable).

A. Take sample prior to the atezolizumab infusion, NOT required during the retreatment period.

B. Take sample prior to the atezolizumab infusion and during the retreatment period.

# 8.4. Analytic Visit Windows for Anti-KTE-C19 Antibody

Table 8-10. Anti-KTE-C19 antibody visit window

| Cohort 1 | Analytic Visit | Baseline | <b>Day 114</b> |
|----------|----------------|----------|----------------|
| | Target Day | Baseline | $114 \pm 7$ |
| | Lab Window | <=-5 | [103, 147] |
| Cohort 2 | Analytic Visit | Baseline | Day 107 |
| | Target Day | Baseline | $107 \pm 7$ |
| | Lab Window | <=-5 | [96, 143] |
| Cohort 3 | Analytic Visit | Baseline | Day 94 |
| | Target Day | Baseline | 94 ± 7 |
| | Lab Window | <=-5 | [78, 143] |

• Baseline antibody samples to be collected prior to start of leukapheresis.

## 8.5. CSF T-cell Analytes

Visits: Screening CSF, Post-CSF, Baseline CSF, Unscheduled CSF

Table 8-11. CSF T-cell analytes

| Number | Name of the analyte (cells/Volume unit) |
|--------|-----------------------------------------------|
| 1 | CD14 (#, gated on CD45+) |
| 2 | CD19 (#, gated on CD45+/66b/14-) |
| 3 | CD3 (#, gated on CD45+/66b/14-) |
| 4 | CD3 CAR+ (#, gated on CD 45+/66b/14-/3+) |
| 5 | CD4 (#, gated of CD45+/66b/14-/3+) |
| 6 | CD4 CAR+ (#, gated on CD45+/66b/14-/3+/4+) |
| 7 | CD45 (#, gated on viable singlets cells) |
| 8 | CD56+CD3- (#, gated on CD45+/66b/14-) |
| 9 | CD56+CD3+(#, gated onCD45+/66b/14-) |
| 10 | CD66b (#, gated on CD45+) |
| 11 | CD8 (#, gated on CD45+/66b/14-/3+) |
| 12 | CD8 CAR+ (#, gated on CD45+/66b/14-/3+/8+) |
| 13 | CSF Volume |
| 14 | Viability (# Total Cells, Gated on Singlets) |
| 15 | Viability (# Viable Cells, Gated on Singlets) |

# 8.6. Using Trapezoidal Rule to Approximate the AUC



AUC 
$$\approx \frac{1}{2}(y_0 + y_1) \cdot \Delta x + \frac{1}{2}(y_1 + y_2) \cdot \Delta x + \frac{1}{2}(y_2 + y_3) \cdot \Delta x + \cdots$$